CLINICAL TRIAL: NCT04730934
Title: Evaluation of the Physical and Emotional Effects of the COVID-19 Pandemic on Fibromyalgia Patients
Brief Title: Effects of the COVID-19 Pandemic on Fibromyalgia Patients
Status: Completed | Type: Observational
Sponsor: Kars State Hospital (Other)
Responsible Party: Principal Investigator, Fatih Bagcier, Medical Doctor, Kars State Hospital
Other Study IDs: 2020/43-01
Record Dates: First submitted 2021-01-28; First posted 2021-01-29 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Fibromyalgia; Chronic Low-back Pain
Keywords: Fibromyalgia; Pandemic; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Perceived Stress Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy population: Healthy individuals aged between 18-65
  Interventions: Other: Perceived stress scale; Other: The drugs used before and during the pandemic, the patient's job status, physical activity conditions, pain status
- Chronic Low Back Pain Group: Patients aged between 18 and 65 and has at least 3 months of low back pain which started before pandemic.
  Interventions: Other: Perceived stress scale; Other: The drugs used before and during the pandemic, the patient's job status, physical activity conditions, pain status
- Fibromyalgia Group: Patients aged between 18 and 65 and has a diagnosis of fibromyalgia for at least 6 months
  Interventions: Other: Perceived stress scale; Other: Fibromyalgia impact questionnaire; Other: The drugs used before and during the pandemic, the patient's job status, physical activity conditions, pain status

INTERVENTIONS:
Other: Perceived stress scale — Perceived stress scale (PSS) : The PSS is a validated 10-item self-report questionnaire which asks individuals to indicate how often they have found their lives unpredictable, uncontrollable, and overloaded in the last month. The higher scores indicating greater perceived stress.
Other: Fibromyalgia impact questionnaire — Fibromyalgia impact questionnaire (FIQ): The FIQ is composed of 10 items. The first item contains 11 questions related to physical functioning - each question is rated on a 4 point Likert type scale. Items 2 and 3 ask the patient to mark the number of days they felt well and the number of days they were unable to work (including housework) because of fibromyalgia symptoms. Items 4 through 10 are horizontal linear scales marked in 10 increments on which the patient rates work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety and depression.
  Groups: Fibromyalgia Group
Other: The drugs used before and during the pandemic, the patient's job status, physical activity conditions, pain status — Drug using: Antidepressant, SNRI, gabapentin, SSRI, myorelaxan, nsaid, paracetamol, pregabalin, tramadol, food supplement.
  Job status: Participants were questioned about their occupational status before and during the pandemic as "I am a housewife", "I quit my job", "I worked from home", "I worked part-time" and "there was no change in my job".
  Physical activity: "I do not have physical activity", "I do my daily work at home", "I do daily walks", "I exercise regularly".
  Pain status: Participants were questioned that their pain conditions before and during the pandemic were "much worse", "worse", "a little bad", "no change", "a little good", " better", It was questioned as "much better".

SUMMARY:
In this study, the effects of the symptoms related to the diseases of patients with fibromyalgia during the COVID-19 pandemic, their limitations in their social and business life, the need for different drugs, stress levels and the effect of the pandemic on the disease activity will be evaluated.

DETAILED DESCRIPTION:
Psychological stress caused by the COVID-19 pandemic may contribute to the severity and duration of physical pain. However, when added to the economic stress due to social isolation, pain may worsen in patients with chronic pain, especially fibromyalgia, prone to anxiety and depression. Due to the fact that many occupational sectors, which concern the whole society, have come to a halt, being obliged to live a sedentary life due to inability to perform their profession may have caused an increase in the body mass index of people. During the pandemic days, our concentration and health services may have shifted from the diseases of our branch to COVID-19 and the branch health services offered may be disrupted. However, the call of the country administrators to stay home and the concept of social isolation caused the routine outpatient clinic follow-ups to be delayed. Lack of sufficient data on how fibromyalgia patients were affected in previous pandemics and the pandemic we are in, the disease levels of the patients in this period, restrictions in their social environment, difficulties in reaching the doctor may have exacerbated the course of the diseases. In this study, the effects of the symptoms related to the diseases of patients with fibromyalgia during the COVID-19 pandemic, their limitations in their social and business life, the need for different drugs, stress levels and the effect of the pandemic on the disease activity will be evaluated. The data to be obtained can be a guiding resource for us in the ongoing pandemic and in the fight against future pandemics due to the mutated genetic structure of the virus.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 65 years
* patients who have low back pain lasting at least 3 months and started before pandemic
* patients diagnosed with fibromyalgia for at least 6 months

Exclusion Criteria:

* patients diagnosed with major depression
* patients who have a history of back surgery, fracture, infection, spinal stenosis
* patients with malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 465 healthy participants, 465 patients with low back pain, 465 patients with fibromyalgia
Sampling Method: Probability Sample
Enrollment: 1360 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Physical activity | 4 weeks
  The physical activities of the participants were evaluated before and during the pandemic with the options "I do not have physical activity", "I do my daily work at home", "I do daily walks", "I exercise regularly".
Occupation conditions | 4 weeks
  Participants were questioned about their occupational status before and during the pandemic as "I am a housewife", "I quit my job", "I worked from home", "I worked part-time" and "there was no change in my job".
General health condition | 4 weeks
  Participants were questioned that their health conditions before and during the pandemic were "much worse", "worse", "a little bad", "no change", "a little good" " better", It was questioned as "much better".
General pain condition | 4 weeks
  Participants were questioned that their pain conditions before and during the pandemic were "much worse", "worse", "a little bad", "no change", "a little good", " better", It was questioned as "much better".
Perceived stress scale | 4 weeks
  Participants were questioned that their stress conditions before and during the pandemic
Fibromyalgia impact questionnaire | 4 weeks
  Fibromyalgia patients were questioned with fibromyalgia impact questionnaire before and during the pandemic

CONTACTS AND LOCATIONS:
Locations (1):
- Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)